CLINICAL TRIAL: NCT07204951
Title: A Double-Blind, Randomized, Control-Arm Clinical Study to Evaluate the Safety and Efficacy of Test Water Flosser in Enhancing Oral Health Among Healthy Adults Having Plaque-Induced Gingivitis and Dental Plaque Accumulation
Brief Title: Clinical Safety and Efficacy Study of Water Flosser in Enhancing Oral Health Among Healthy Adults Having Plaque-induced Gingivitis and Dental Plaque Accumulation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NovoBliss Research Pvt Ltd (Other)
Collaborators: GuruNanda LLC (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: NB250034-GN_1.0_23Sep25
Record Dates: First submitted 2025-09-24; First posted 2025-10-03 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Plaque Induced Gingivitis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Gurunanda - Water Flosser (Experimental): Mode of Usage: Follow the below listed steps for product usage post brushing of teeth.
  1. Fill - Add water to the tank of the Flosser
  2. Insert - Add the tip to the flosser
  3. Select - Choose the level of pressure
  4. Floss - Guide the stream between your teeth and along the gumline
  5. Clean - After use, insert the tip in the water tank and sanitize Frequency: Use twice a day after brushing. Route of administration: Topical - Oral Storage Condition: Store in a cool, dry place, away from direct sunlight, and do not submerge in water.
  Interventions: Device: Gurunanda - Water Flosser
- No water Flossing (Experimental)
  Interventions: Other: No water Flossing

INTERVENTIONS:
Device: Gurunanda - Water Flosser — Mode of Usage: Follow the below listed steps for product usage post brushing of teeth.
  1. Fill - Add water to the tank of the Flosser
  2. Insert - Add the tip to the flosser
  3. Select - Choose the level of pressure
  4. Floss - Guide the stream between your teeth and along the gumline
  5. Clean - After use, insert the tip in the water tank and sanitize Frequency: Use twice a day after brushing. Route of administration: Topical - Oral Storage Condition: Store in a cool, dry place, away from direct sunlight, and do not submerge in water.
  Arms: Gurunanda - Water Flosser
Other: No water Flossing — No water Flossing
  Arms: No water Flossing

SUMMARY:
This is a double-blind, randomized, control-arm clinical study to evaluate safety and efficacy of test water flosser in enhancing oral health among healthy adults having plaque-induced gingivitis and dental plaque accumulation.

DETAILED DESCRIPTION:
A total of 64 subjects, including males and non-pregnant, non-lactating females aged between 18 and 65 years (inclusive) with mild to moderate plaque-induced gingivitis will be enrolled to ensure 60 subjects (30 subjects/arm) to complete the study. Subjects will be screened as per the inclusion & exclusion criteria after obtaining written informed consent.

There will be a total of 3 visits during the study. The duration of the study will be 30 Days (±2 Days) from the enrolment.

Visit 01(Day 01): Screening, ICD obtained, Enrolment, Baseline Evaluation, Product Usage & T30mins Evaluations.

Visit 02 [Day 15 ((±2 Days)]: Test Product Usage Period, Oral Assessments Visit 03[Day 30 (±2 Days)]: Oral Assessments, End of Study.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 to 65 years (both inclusive) old at the time of consent.
2. Sex: Healthy adult males and non-pregnant/non-lactating females.
3. Females of childbearing potential have a self-reported negative urine pregnancy test at the time of the screening visit and agree to follow an accepted method of birth control for the duration of the study such as condoms, foams, jellies, diaphragm, intrauterine device etc.
4. Subjects are generally in good general health as determined from recent medical history.
5. Subjects with mild to moderate gingivitis and good oral health, without hard or soft tissue lesions, with moderate gingivitis characterized by more than 30% bleeding sites and probing depths of ≤3 mm without attachment loss.
6. Anterior teeth without restorations.
7. No dental treatments being performed before or during the study period.
8. Possessing at least 20 permanent teeth (excluding the third molars) and 5 evaluable teeth in each quadrant.
9. Subjects who agree to discontinue the use of over-the-counter any teeth products throughout the trial except for the ADA-approved toothbrush and toothpaste provided during the study.
10. Subjects who agree to refrain from the use of any other type of floss or similar dental product during the study.
11. Agree not to participate in any other oral/dental product studies during the trial.
12. Agree to return for all scheduled visits and follow study procedures.
13. Subjects who are willing to complete all study procedures including study-related questionnaires and comply with study requirements.

Exclusion Criteria:

1. Subjects who are undergoing treatment for gingivitis, caries, dental plaque and sensitivity.
2. Subjects are present with fixed orthodontic appliances on the facial surfaces of the maxillary arch.
3. Subjects have dental crowns, veneers or composite restorations on gradable maxillary anterior teeth (canine to canine) or mandibular anterior teeth.
4. Subjects have any oral pathologies or gross neglect of home care requiring prompt treatment, including periodontal disease, as evidenced by purulent exudate, tooth mobility, and/or other signs indicating that the integrity of the data collected for that subject might be compromised.
5. Subjects are present with any pre-existing oral or medical condition that the Investigator/designee determines may place the subject at increased health risk from study participation.
6. Suffering from untreated dental caries, mucosal lesions, oral tumors or severe systemic diseases that may affect periodontal diseases.
7. Subjects have any known allergies to over-the-counter oral hygiene/products.
8. Subjects have any known allergies to the trial product ingredients.
9. The subject must have participated in a clinical study with oral care or oral hygiene within 4 weeks before the screening visit of this study.
10. Any other condition which could warrant exclusion from the study, as per the Investigator's discretion
11. Subjects who smoke and are pan eaters.
12. Subjects with hypersensitive teeth.
13. Subjects having chipped teeth and defective restorations.
14. Subjects having deep periodontal pockets.
15. Subjects having bridgework in their teeth and dentures which interrupt during evaluation.
16. Subjects undergoing treatment with antibiotics, anti-inflammatory, anticonvulsants, anti-histaminic, anti-depressant, anti-histaminic, sedatives, tranquilizers or daily analgesic drugs.
17. Subjects having uncontrolled metabolic disease.
18. Subjects' overexposure to acidic by dietary and environment exposure.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2025-11-13 (Estimated); Primary Completion 2025-11-13 (Estimated); Study Completion 2025-12-06 (Estimated)

PRIMARY OUTCOMES:
To assess the effectiveness of the test product in terms of change in plaque deposition | Before and after usage of test product at T30 mins on Day 01, Day 15 (±2 days), and Day 30 (±2 days)
  By using Turesky Modification of the Quigley-Hein Index by Dentist or Dentist trained evaluator.
To assess the effectiveness of the test product in terms of change in plaque induced gingivitis | Before and after usage of test product at T30 mins on Day 01, Day 15 (±2 days), and Day 30 (±2 days)
  By using Loe & Silness Gingival Index by Dentist or Dentist trained evaluator.

SECONDARY OUTCOMES:
To assess the improvement in product perception questionnaire | Baseline prior to usage of test product and on Day 01, Day 15 (±2 days), and Day 30 (±2 days)
  Quality of life questionnaire through 5-point Likert scale to evaluate the changes in plaque formation

OTHER OUTCOMES:
Safety assessment by examined of oral soft tissues (tongue, hard and soft palate, gingivae, mucobuccal folds, inner cheeks, sublingual areas) and hard tissues, including dental restorations. | At baseline Day 01 (±2 days), Day 15 (±2 days), and Day 30 (±2 days)
  Safety will be assessed by a dentist or dentist-trained evaluator. Findings will be categorized as normal or abnormal and analyzed using an appropriate nonparametric test.

CONTACTS AND LOCATIONS:
Overall Officials: Nayan Patel, Study Director — NovoBliss Research Pvt Ltd

IPD SHARING:
Plan to Share IPD: No